CLINICAL TRIAL: NCT03115255
Title: Serum Concentrations of Vascular Endothelial Growth Factor in Infants Treated With Ranibizumab for Retinopathy of Prematurity
Brief Title: Serum Vascular Endothelial Growth Factor in Infants With Intravitreal Ranibizumab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: XH-17-004
Record Dates: First submitted 2017-03-27; First posted 2017-04-14 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-04

CONDITIONS: Infant, Premature, Diseases
Keywords: retinopathy of prematurity; ranibizumab; vascular endothelial growth factor
MeSH Terms: conditions — Infant, Premature, Diseases; Retinopathy of Prematurity | interventions — Ranibizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- serum VEGF level (Experimental): Serum samples are collected 1 day before and 1 day, 3 days, 1 week after intravitreal ranibizumab
  Interventions: Drug: intravitreal ranibizumab

INTERVENTIONS:
Drug: intravitreal ranibizumab — 0.25 mg intravitreal ranibizumab to either 1 eye (unilateral cases) or both eyes (bilateral cases)
  Other Names: lucentis

SUMMARY:
To determine the serum concentrations of ranibizumab and vascular endothelial growth factor (VEGF) in infants with retinopathy of prematurity (ROP) who received intravitreal ranibizumab

DETAILED DESCRIPTION:
Infants with ROP are studied. They received 0.25 mg or 0.5 mg of intravitreal ranibizumab to either 1 eye (unilateral cases) or both eyes (bilateral cases) with vascularly active ROP. Serum samples are collected 1 day before and 1 day, 3 days, 1 week after intravitreal ranibizumab. The serum concentrations of ranibizumab and VEGF are measured by enzyme-linked immunosorbent assay, and the changes of the serum VEGF levels are determined.

ELIGIBILITY:
Inclusion Criteria:

* Infants with vascularly active ROP
* intravitreal ranibizumab

Exclusion Criteria:

* already accepted laser therapy

Ages: 4 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The effect of intravitreal ranibizumab on serum VEGF level | 1 day before and 1 day, 3 days, 1 week after intravitreal ranibizumab
  the changes of the serum VEGF levels

SECONDARY OUTCOMES:
The effect of intravitreal ranibizumab on weight | corrected age of six month
  measure weight of the infants
The effect of intravitreal ranibizumab on height | corrected age of six month
  measure height of the infants
The effect of intravitreal ranibizumab on neurologic development | corrected age of six month
  Gesell development diagnosis scale

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Xia, MD. PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No